CLINICAL TRIAL: NCT06464809
Title: Treatment Effects of Transcutaneous Electrical Nerve Stimulation and Kinesio Taping on Hand Functions for Patients With Carpal Tunnel Syndrome
Brief Title: Treatment Intervention of Patients With Carpal Tunnel Syndrome (CTS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Wei-Hsien Hong, Associate Professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH103-REC3-072
Record Dates: First submitted 2024-06-04; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome; home-based treatment program; kinesio taping; paresthesia; thenar eminence
MeSH Terms: conditions — Carpal Tunnel Syndrome; Paresthesia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This was a prospective, randomized-controlled trial.
Who Masked: Participant
Masking Description: The participants who met the inclusion criteria were randomized into one of two treatment groups: KT group and TENS group. Participants were blinded to the treatments used in the other group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesio taping (KT) group (Experimental): Three precut KT I strips with a width of 5 cm were used. The first strip is applied with the subject's wrist in fully extended hand position. Middle and ring fingers through the holes with the base of the tape as anchored to the knuckles, and then the tape was applied with 15%-25% tension covering the palm and the wrist, and the remainder of the tape without any tension from the wrist up to the forearm. The same process is repeated for the second I-strip, which was applied from the dorsum of the hand to wrist while the wrist in a downward flexed position. The final strip was applied to the carpal tunnel region with 25%-35% tension.
  Interventions: Other: kinesio taping (KT)
- transcutaneous electrical nerve stimulation (TENS) group (Active Comparator): A portable TENS unit (Gem-Stim, Gemore Technology Co., LTD. Taiwan) was used, and delivered a bi-phasic symmetric waveform at a continuous frequency of 100 Hz and phase duration of 200 µsec. The intensity was gradually adjusted up to a strong but comfortable l level, as reported by the subject. Two electrodes were placed 2 cm apart, respectively attached to the carpal ligament of the affected side and the proximal end along the direction of the median nerve.
  Interventions: Other: kinesio taping (KT)

INTERVENTIONS:
Other: kinesio taping (KT)
  Other Names: transcutaneous electrical nerve stimulation (TENS)

SUMMARY:
The purpose of this study was to investigate the effectiveness of KT versus TENS combining self-myofascial stretching in treatment of CTS through clinical, functional assessment and sensory measurements.

Primary hypothesis The KT group has a more substantial improvement in hand grip, pain relief, enhancing proprioceptive sensitivity and dexterity compare to the TENS group. treatment program,

DETAILED DESCRIPTION:
Objective: To compare the effectiveness of a home-based treatment program involving Kinesio taping (KT) or transcutaneous electrical nerve stimulation (TENS) among carpal tunnel syndrome (CTS) patients.

Methods:

30 participants with CTS were enrolled, age range, 30 to 60 years. The participants who met the inclusion criteria were randomized into one of two treatment groups: KT group and TENS group. Participants were blinded to the treatments used in the other group.

Patients with CTS received aforementioned treatments compared with reliable qualitative and quantitative evaluation tools before and after 4-week treatment, as well as at a additional 4-week follow-up. The main parameters include the Symptom Severity Scale (SSS) and Functional Status Scale (FSS), hand grip and key pinch strengths, two-point discrimination (2PD), Modified Moberg pick-up test (MMPUT), and Pain assessment (visual analog scale, VAS).

ELIGIBILITY:
Inclusion Criteria:

* numbness and tingling in the median nerve territory of the hand.
* nocturnal paresthesia.
* induction test (Tinel's sign and Phalen's test) showing a positive finding.,
* is defined as mild and moderate CTS according to nerve conduction studies (NCSs).

Exclusion Criteria:

* is defined severe CTS symptoms.
* are currently pregnant or have any secondary entrapment neuropathy (e.g., diabetes, inflammatory arthritis, hypothyroidism, previous wrist trauma).
* cervical radiculopathy or polyneuropathy.
* previous history of carpal tunnel decompression surgery.
* corticosteroid injection into the carpal tunnel.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09-24 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
The SSS and FSS of the Boston Carpal Tunnel Questionnaire (BCTQ) | pre-intervention, 4-week intervention, and 4-week follow-up.
  Assess symptoms and functional status. The SSS subscale includes 11 items assessing pain, paresthesia, numbness, weakness, nocturnal symptoms and over-all functional status. The FSS subscale includes 8 items assessing the hand function during common daily activities. Each item is scored on a 5-point scale (1-5), from 1(no symptoms) to 5 (the worst symptoms) for SSS, and from 1 (no difficulty) to 5 (cannot perform the activity at all) for FSS. The overall SSS and FSS scores are calculated as the mean of the scores for 11 and 8 individual items respectively, such that the higher the score obtained, the worse the SSS or FSS.
Hand grip and key pinch strengths | pre-intervention, 4-week intervention, and 4-week follow-up.
  pinch strength included palmar, three-jaw chuck, tip, and lateral pinches.
Two-point discrimination (2PD) | pre-intervention, 4-week intervention, and 4-week follow-up.
  cutaneous sensory perception threshold. The larger the value of distance, the worse the sensory ability.
Modified Moberg pick-up test (MMPUT) | pre-intervention, 4-week intervention, and 4-week follow-up.
  hand dexterity. The shorter the time, the more dexterity the hand.
The visual analog scale (VAS) | pre-intervention, 4-week intervention, and 4-week follow-up.
  pain measurement. 100 mm straight line, with 0 mm on the far left and 100 mm on the far right, 0 mm positions It is not painful, and 100 mm is extremely painful.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Hsien Hong, PhD, Principal Investigator — China Medical University, Taiwan
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No